CLINICAL TRIAL: NCT04700358
Title: Identification and Characterization of Antibacterial Antibodies in Sera of Patients With Cystic Fibrosis
Brief Title: Characterization of Antibacterial Antibodies in Patients With Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Alexander Simonis, MD, University of Cologne
Other Study IDs: 20-1287_1
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Cystic Fibrosis; Neutralizing Antibodies
MeSH Terms: conditions — Cystic Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Serum and PBMCs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Cystic Fibrosis: Patients with pulmonary Cystic Fibrosis with or without bacterial colonization
  Interventions: Other: Blood sampling
- Control group: Healthy age- and sex-matched controls including healthy individuals and patients with acute or chronic bacterial infections
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Screening: Blood sampling of 15 ml whole blood
  B cell isolation: Blood sampling of max. 400 ml whole blood or 6% of the total blood volume (♀ 65 ∓ 10 ml/kg; ♂ 77 ∓ 10 ml/kg)

SUMMARY:
Most of the cystic fibrosis (CF) patients are or have been pulmonary colonized with bacteria such as Pseudomonas aeruginosa or Staphylococcus aureus. Aim of this study is to detect virulence factor neutralizing antibodies in the sera of the study population followed by B cell repertoire analyses to design B cell-derived neutralizing monoclonal antibodies. The functionality of neutralizing antibodies rests on inhibition of virulence factors by binding of crucial epitopes rather than merely the induction of opsonization. Focusing on patients with bacterial colonization/chronic infections or a history of an acute infection in the past, will increase the likelihood for identification of serum with neutralizing activity as in vivo antigen contact is a prerequisite for antibody development and maturation. Since virulence factors are essential for infection, dissemination and tissue damage, inhibition of these factors by developed neutralizing antibodies might contribute to a favorable outcome of life-threatening infections.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to give consent
* Normal vital signs including:
* Blood pressure systolic value 150 - 100 mmHg, diastolic value < 90 mmHg
* Respiratory rate < 20/min
* Oxygen saturation >92%
* Heart rate 50 - 110/min
* Body temperature <38°C

Exclusion Criteria:

* Cytopenia (leukocytes < 1.500/µl, thrombocytes < 50.000/µl, Hemoglobin < 12 g/dl)
* Heart disease or pulmonary hypertension
* Body weight <50 kg (exclusion of blood sampling for B cell isolation)
* Blood donation, larger blood loss and/or major surgery in the last 8 (male) or 12 (female) weeks
* Any decline of the general state of health in the last 3 month including weight loss > 2kg, pulmonal exacerbation or increased impairment of pulmonary function (FEV1 < 50%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the University Hospital Cologne
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of antibacterial antibodies | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Silke van Koningsbruggen-Rietschel, MD, PhD, Study Director — University Hospital Cologne; Jan Rybniker, MD, PhD, Study Director — University Hospital Cologne
Locations (1):
- CF Study Center, University Hospital Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided